CLINICAL TRIAL: NCT03258736
Title: Comparison of Caudal Block and Ultrasound Guided Ilioinguinal/Iliohypogastric Block for Bilateral Inguinal Surgery in Pediatric Patient: A Prospective Randomized Trial
Brief Title: Caudal Block Versus Ultrasound Guided Ilioinguinal/Iliohypogastric Block in Pediatric Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayse Cigdem Tutuncu, assoc prof, Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 604.01/02-7626
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-04

CONDITIONS: Surgery
Keywords: pediatric, inguinal hernia, caudal, ilioinguinal/ilioihypogastric
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block (Other): Caudal block Marcaine
  Interventions: Procedure: inguinal hernia surgery
- ilionguinal/iliohypogastric block (Other): ilionguinal/iliohypogastric block Marcaine
  Interventions: Procedure: inguinal hernia surgery

INTERVENTIONS:
Procedure: inguinal hernia surgery — repair of inguinal hernia

SUMMARY:
The caudal block is the most common technique for inguinal surgery. Increased use of ultrasound in regional analgesia techniques has been improved the practise of the peripheral nerve blocks. Ilioinguinal and iliohypogastric nerve blocks are possible to alternative methods to the central blocks. The aim of this study is to compare analgesic efficiency of caudal block and ultrasound guided Ilioinguinal and iliohypogastric nerve blocks for bilateral inguinal hernia in pediatric patients

DETAILED DESCRIPTION:
In this prospective randomized study, pediatric patients between 1- 10 years old who were scheduled to bilateral inguinal hernia surgery wil be enrolled the study. The patients wil randomly assign to receive an ultrasound-guided Ilioinguinal/iliohypogastric block group or caudal block group Ilioinguinal/iliohypogastric block was performed with 2 mg/kg bupivacaine as 0.25 % and total volum wil be divided equally for each side, Caudal block wil performe with bupivacaine 2 mg/kg as 0.2%. Supplemental analgesia will consist of as requred intraoperative remifentanyl, for recovery unit rescue tramadol, as requred at home ibuprofen. Patients wil be evaluated in the recovery unit for analgesia with FLACC pain scale, analgesic requirement, complications and parental satisfaction. Parents will be also called for analgesia and satisfaction after discharge of the patients in first 24 hours. The evaluation will be performed by a researcher whom does not know which participants belong to the caudal or ilioinguinal/iliohypogastric nerve block group

ELIGIBILITY:
Inclusion Criteria:1- 10 year- old who were scheduled to bilateral inguinal hernia surgery -

Exclusion Criteria: Patients with neurological disoder, reoperation for inguinal hernia surgery, coagulation disorder

-

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Analgesic requirements | up to 24 hours
  FLACC score

SECONDARY OUTCOMES:
Postoperative complications | up to 24 hours
  Bromage scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa Medical Faculty, Istanbul, Cerrahpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Availabe from the authors